## **Consent Form**

Neuroepidemiology Unit Centre for Epidemiology and Biostatistics Melbourne School of Population and Global Health Faculty of Medicine, Dentistry and Health Sciences The University of Melbourne



## **Project:** An Online Educational Course for people with Multiple Sclerosis: A randomised controlled trial of course effectiveness

**Responsible Researcher:** Dr Sandra Neate, Head of Neuroepidemiology Unit, senior

research fellow

**Additional Researchers:** Dr Jeanette Reece, investigator, epidemiologist; Mr. William Bevens, research assistant, PhD candidate; Professor George Jelinek, investigator; Dr Nupur Nag, investigator; Ms Maggie Yu, research assistant, data manager; Professor Kathleen Gray, investigator; Dr Steve Simpson-Yap, investigator, biostatistician; Dr Pia Jelinek, investigator

## Name of Participant:

- 1. I consent to participate in this project, the details of which have been explained to me, and I have been provided with a written plain language statement to keep.
- 2. I understand that the purpose of this research is to investigate the effectiveness of the two online courses (the Multiple Sclerosis Online intervention course and the Multiple Sclerosis Online standard-care course) in improving physical and mental health outcomes in people with MS.
- 3. I understand that my participation in this project is for research purposes only.
- 4. I acknowledge that the possible effects of participating in this research project have been explained to my satisfaction.
- 5. In this project I will be required to:
  - Complete a baseline survey related to my lifestyle and health
  - Complete the Multiple Sclerosis Online course related to diet, exercise, sunlight and vitamin D, stress reduction and other information about multiple sclerosis. The course comprises 8 modules of approximately one hour each and the modules must be completed within a six-week period.
  - Complete a survey related to my lifestyle and health at 6 months, 1 year and 2.5 years after completing the Online course.

Ethics ID Number: 22140 Project Start Date: 1 November, 2021 Version: 1

- One month and 12 months after completing the Online course, I may be invited to participate in a 30-60 minute phone or internet interview about my experience of the Online course and any impact it may have had on me. However, I have the option to decline participating in these interviews.
- 6. I understand if I agree to participate in any interviews, these interviews will be audio-taped and transcribed by voice recognition software.
- 7. I understand that my participation is voluntary and that I am free to withdraw from this project anytime without explanation or prejudice and to withdraw any unprocessed data that I have provided.
- 8. I understand that the data from this research will be stored indefinitely at the University of Melbourne.
- 9. I have been informed that the confidentiality of the information I provide will be safeguarded subject to any legal requirements; my data will be password protected and accessible only by the named researchers.
- 10. This form is provided for your information you are not expected to sign or return this form. Your consent to participate is implied when you click on the link to agree to participate in the baseline survey.

| Participant Consent: |
|-------------------------------------------------|
| Please tick to give your consent to participate |